CLINICAL TRIAL: NCT06448884
Title: Accuracy of the Caries Risk Assessment of International Caries Classification and Management System (ICCMS) Versus Simplified Cariogram in the Egyptian Young Adult Population
Brief Title: Accuracy of ICCMS Versus Simplified Cariogram
Status: Not yet recruiting | Type: Observational
Sponsor: Kirolos Hisham Nadi Sedek (Other)
Responsible Party: Sponsor-Investigator, Kirolos Hisham Nadi Sedek, Principal Investigator, Cairo University
Organization: Cairo University (Other)
Other Study IDs: 29607210104331
Record Dates: First submitted 2024-05-29; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Caries,Dental
Keywords: Risk; Validity; Cariogram; ICCMS
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to compare the validity of the caries risk assessment regarding the comprehensive ICCMs Caries risk and likelihood matrix versus the simplified Cariogram aiming to see if there is a significant difference in the caries risk levels between both models.

DETAILED DESCRIPTION:
The simplified Cariogram has been already established as a simple computerised efficient way to categorise patients according to their risk of developing new lesions. However, since then, more comprehensive ways such as the ICCMS have risen. Such comprehensive models require much more data to be entered and more time for the assessment to be complete.

This study aims to test whether there is a significant difference between the validity of both models that would justify the extra time, effort, and recordings that have to be taken for the ICCMS.

ELIGIBILITY:
Inclusion Criteria:

* Age ranging from 18 to 29 years.
* The presence of dental caries or restoration.

Exclusion Criteria:

* Patients with no caries.
* Patients diagnosed of psychiatric disease.
* Patients not willing to be part of the study or ones who refuse to sign the informed consent.

Ages: 18 Years to 29 Years | Sex: All
Age Groups: Adult
Study Population: Young Adult Egyptians
Sampling Method: Non-Probability Sample
Enrollment: 323 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Validity | At baseline Immediately after collecting the data.
  Measured in terms of sensitivity and specificity between the data set of the intervention and the comparator using ROC analysis.
  There will be no need for follow up records as we are comparing 2 Patient Caries risk classification models. The models determine the Patient's risk category immediately after the required data is inserted into them.

SECONDARY OUTCOMES:
Reproducibility | At baseline Immediately after collecting the data.
  It will be measured based on the level of agreement between the results using KAPPA analysis. There will be no need for follow up records as we are comparing 2 Patient Caries risk classification models. The models determine the Patient's risk category immediately after the required data is inserted into them.